CLINICAL TRIAL: NCT05741892
Title: 3D Planned Surgery of Acute Fractures Performed With 3D Guides Printed at the Point of Care - a Prospective Case Series
Brief Title: 3D Planned Surgery of Acute Fractures Performed With 3D Guides Printed at the Point of Care
Acronym: 3DFRG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5364
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Fracture Tibia; Fracture Femur; Fracture, Comminuted
Keywords: Femur; Tibia; Comminuted fracture; 3D printing; personalized medicine
MeSH Terms: conditions — Tibial Fractures; Femoral Fractures; Fractures, Comminuted

STUDY DESIGN:
Intervention Model Description: Prospective case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D fracture reposition guide group (Experimental): Comminuted tibial- or/and femur shaft fractures will be treated using 3D printed patient-specific repositions guides.
  Interventions: Device: Fracture reposition with 3D printed patient specific repositions guides

INTERVENTIONS:
Device: Fracture reposition with 3D printed patient specific repositions guides — Comminuted tibial- or/and femur shaft fractures will be treated using 3D printed patient-specific repositions guides.

SUMMARY:
The aim of the study is to assess the accuracy of fracture reduction performed with surgical guides designed and 3D printed at the point of care in comminuted fractures of femur- and tibia-shaft.

DETAILED DESCRIPTION:
The 3D planning of surgeries and their execution with 3D printed templates adapted to the individual patient is an established procedure for elective surgeries such as corrective osteotomies for mal-united fractures. Currently, the planning and production of 3D templates are performed mainly by external companies. The duration until delivery usually exceeds four weeks. Therefore, it is not possible to use them in acute cases (e.g. acute fractures) that need to be treated surgically within a few days.

The most frequent postoperative deformity in long bone shaft fractures is malrotation. In femoral fractures, clinically relevant rotational errors (>15°) occur in up to 40% of cases after surgical treatment, which either results in a poor clinical outcome or requires revision surgery. In tibial diaphyseal fractures, up to 50% of rotational errors have been reported. The higher the degree of comminution the higher the chances of malrotation postoperatively. Due to the comminuted situation, no reliable bony references exist intraoperatively and the surgeon can only estimate the correct length, axis and, rotation based on the contralateral leg. This ultimately leads to a high number of revision surgeries or poor outcomes. Porcine and human cadaveric feasibility studies conducted by the study team utilizing site 3D planned and printed reduction guides showed excellent accuracy of fracture reduction.

This project aims to apply this technique to the clinical setting by conducting a clinical study. The accuracy of 3D planned surgery performed with surgical guides designed and printed at the point of care will be assessed and the complication rate will be compared to the known literature.

It was hypothesized that the mean deviation between the measured postoperative rotational alignment and planned rotation alignment in patients treated for comminuted fractures of femur- and tibia-shaft treated using 3D printed reposition guides will be less than 5°. Additionally, it was hypothesized that the rate of clinically relevant deviations between postoperative rotational alignment (e.g. 15°) and planned rotation in patients treated for comminuted fractures of femur- and tibia-shaft treated using 3D printed reposition guides will be less than 10%.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 99 years
* Comminuted shaft fracture of tibia or femur
* Intact contralateral tibia or femur
* Patient willing to participate and sign the informed consent
* Clear indication of surgical treatment

Exclusion criteria:

* Refusal to sign the informed consent
* Abnormal contralateral bony anatomy (previous surgeries, poliomyelitis, previous injury, implants)
* Pregnancy
* Acute tumor or previous tumor disease
* Acute infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Rotational deviation (Axial plane deviation) in degree | Between 1 to 7 days postoperative, depending on the patients status
  Planned rotational alignment versus postoperative rotational alignment.

SECONDARY OUTCOMES:
Length deviation in mm | Between 1 to 7 days postoperative, depending on the patients status
  Planed length versus postoperative length
Frontal plane deviation in degree | Between 1 to 7 days postoperative, depending on the patients status
  Planned varus/valgus alignment versus postoperative varus/valgus alignment
Sagittal plane deviation in degree | Between 1 to 7 days postoperative, depending on the patients status
  Planned flexion/extension of the proximal and distal fracture fragments compared to the postoperative position.

CONTACTS AND LOCATIONS:
Overall Officials: Hecker Andreas, MD, Principal Investigator — Universitätsklinik für Orthopädische Chirurgie und Traumatologie
Locations (1):
- Universitätsklinik für Orthopädische Chirurgie und Traumatologie, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No